CLINICAL TRIAL: NCT05357755
Title: A Phase 2a Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of an Oral Tablet Formulation of JNJ-77242113 for the Treatment of Moderate-to-Severe Plaque Psoriasis
Brief Title: A Study of JNJ-77242113 for the Treatment of Moderate-to-Severe Plaque Psoriasis
Acronym: SUMMIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109193; 2021-005987-23 (EudraCT Number); 77242113PSO2003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: JNJ-77242113 Dose 1 (Experimental): Participants will receive JNJ-77242113 Dose 1 as delayed release tablets orally once daily from Week 0 through Week 16.
  Interventions: Drug: JNJ-77242113
- Group 2: JNJ-77242113 Dose 2 (Experimental): Participants will receive JNJ-77242113 Dose 2 as delayed release tablets orally once daily from Week 0 through Week 16.
  Interventions: Drug: JNJ-77242113
- Group 3: Placebo (Placebo Comparator): Participants will receive oral dose of matching placebo once daily from Week 0 through Week 16.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-77242113 — JNJ-77242113 will be administered orally as delayed release tablets.
  Other Names: PN-21235,; PN-235
  Arms: Group 1: JNJ-77242113 Dose 1; Group 2: JNJ-77242113 Dose 2
Drug: Placebo — Matching placebo will be administered orally as delayed release tablets.
  Arms: Group 3: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy of an oral tablet formulation of JNJ-77242113 compared with placebo in participants with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
The population of people living with moderate to severe psoriasis is approximately 3.5 billion who are mostly managed with topical and conventional therapies. JNJ-77242113, investigational drug, targets the immune responses in the body and skin which impacts diseases, such as psoriasis and psoriatic arthritis and this study evaluates JNJ-77242113 as options of advanced therapies in moderate to severe plaque psoriasis. The hypothesis of this study is that an oral tablet formulation of JNJ-77242113 will result in superior efficacy compared with placebo as determined by the percentage of participants achieving Psoriasis Area and Severity Index (PASI) 75 (greater than or equal to [>=] 75 percentage [%] improvement in PASI) (PASI 75) response at Week 16. The total duration of this study is up to 24 weeks which includes a screening period of less than or equal to (<=) 4 weeks, a 16-week placebo- controlled treatment period, and a follow-up visit approximately 4 weeks after the last administration of study intervention. Safety assessments include adverse events (AEs) monitoring, clinical safety laboratory assessments, electrocardiograms (ECGs), vital signs, physical examinations, concomitant medication monitoring, pregnancy testing, Columbia Suicide Severity Rating Scale (C-SSRS) and tuberculosis evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of plaque psoriasis, with or without psoriatic arthritis, for at least 26 weeks prior to the first administration of study intervention
* Participant has a total Body Surface Area (BSA) greater than or equal to (>=) 10 percentage (%) at screening and baseline
* Participant has a total Psoriasis Area and Severity Index (PASI) >= 12 at screening and baseline
* Participant has a total Investigator's Global Assessment (IGA) >= 3 at screening and baseline
* Participant be a candidate for phototherapy or systemic treatment for plaque psoriasis

Exclusion Criteria:

* Participant has a nonplaque form of psoriasis (for example, erythrodermic, guttate, or pustular)
* Participant has current drug-induced psoriasis (for example, a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
* Participant have previously received any other therapeutic agent directly targeted to interleukin 23 (including but not limited to guselkumab, tildrakizumab, or risankizumab)
* Participant has received any therapeutic agent directly targeted to interleukin 17 (IL-17), interleukin 17 receptor (IL-17R) or interleukin 12/23 (IL-12/23) (including but not limited to secukinumab, ixekizumab, brodalumab, or ustekinumab) or has received biological therapy targeting tumor necrosis factor (TNF) (including, but not limited to adalimumab, infliximab, or etanercept) within 12 weeks or 5 half-lives, whichever is longer, of the first administration of study intervention
* Participant has received proton pump inhibitors (including but not limited to omeprazole, esomeprazole, lansoprazole, rabeprazole, pantoprazole, dexlansoprazole, or zegerid) within 1 week of first administration of study intervention

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Psoriasis Area Severity Index (PASI) 75 Score at Week 16 | Week 16
  Percentage of participants achieving PASI 75 score (greater than or equal to [>=] 75 percentage [%] improvement from baseline in PASI) at Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: head, trunk, upper, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to Week 24
  An adverse event is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the intervention.
Number of Participants with Serious Adverse Events (SAEs) | Up to Week 24
  SAE is an adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.
Change from Baseline in PASI Total Score at Week 16 | Baseline and Week 16
  Change from baseline in PASI total score at Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: head, trunk, upper, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percentage of Participants Achieving PASI 90 Score at Week 16 | Week 16
  Percentage of participants achieving PASI 90 score (>=90% improvement from baseline in PASI) at Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: head, trunk, upper, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percentage of Participants Achieving PASI 100 Score at Week 16 | Week 16
  Percentage of participants achieving PASI 100 score (100% improvement from baseline in PASI) at Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: head, trunk, upper, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percentage of Participants Achieving an Investigator's Global Assessment (IGA) Score of Cleared (0) or Minimal (1) at Week 16 | Week 16
  Percentage of participants achieving an IGA score of cleared (0) or minimal (1) at Week 16 will be reported. The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Percentage of Participants Achieving an IGA Score of Cleared (0) at Week 16 | Week 16
  Percentage of participants achieving an IGA score of cleared (0) at Week 16 will be reported. The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Change from Baseline in Body Surface Area (BSA) at Week 16 | Baseline and Week 16
  Change from baseline in BSA at Week 16 will be reported. BSA is a commonly used measure of extent of skin disease. It is defined as the percentage of surface area of the body involved with the condition being assessed (that is, plaque psoriasis).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (34):
- United States (12):
  - Stoll Dermatology, Beverly Hills, California
  - Northshore University Healthsystem, Skokie, Illinois
  - Epiphany Dermatology of Kansas, LLC, Overland Park, Kansas
  - Dermatology Specialists, Louisville, Kentucky
  - Lawrence J Green MD LLC, Rockville, Maryland
  - ActivMed Practices and Research, Beverly, Massachusetts
  - ActivMed Practices and Research, Portsmouth, New Hampshire
  - Windsor Dermatology, PC, East Windsor, New Jersey
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - The Pennsylvania Centre for Dermatology, LLC, Exton, Pennsylvania
  - Health Concepts, Rapid City, South Dakota
  - Arlington Center for Dermatology, Arlington, Texas
- Canada (5):
  - Dermatology Research Institute Inc, Calgary, Alberta
  - The Guenther Dermatology Research Centre, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - DermEdge Research, Mississauga, Ontario
  - Toronto Research Centre, Toronto, Ontario
- France (4):
  - CHRU Brest - Hopital Morvan, Brest
  - CHU de Grenoble Hopital Albert Michallon, La Tronche
  - CHU de Nice Hopital de l Archet, Nice
  - Polyclinique de Courlancy, Reims
- Germany (7):
  - Hautarztpraxis, Bramsche
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden
  - Privatpraxis Dr. Hilton & Partner, Düsseldorf
  - Universitatsklinikum Frankfurt, Frankfurt am Main
  - Universitatsklinikum Schleswig Holstein Campus Lubeck, Lübeck
  - Universitatsklinikum Munster, Münster
  - Universitaetsmedizin Rostock, Rostock
- Poland (3):
  - Specderm Poznanska sp j, Bialystok
  - Specjalistyczny gabinet dermatologiczny Aplikacyjno Badawczy Marek Brzewski Pawel Brzewski Spolka Cywilna, Krakow
  - Centrum Terapii Wspolczesnej J M Jasnorzewska Spolka Komandytowo Akcyjna, Lodz
- Spain (3):
  - Hosp. Univ. de Cruces, Barakaldo
  - Hosp. Univ. San Cecilio, Granada
  - Hosp. Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency